CLINICAL TRIAL: NCT00864396
Title: Twice Daily Prevacid for the Treatment of Laryngopharyngeal Reflux: A Double-Blind, Placebo Controlled, Randomized Clinical Trial
Brief Title: Twice Daily Prevacid for the Treatment of Laryngopharyngeal Reflux
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200513298
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2009-03

CONDITIONS: Laryngopharyngeal Reflux
Keywords: Laryngopharyngeal reflux; Gastroesophageal reflux disease; GERD
MeSH Terms: conditions — Laryngopharyngeal Reflux; Gastroesophageal Reflux | interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevacid (Experimental)
  Interventions: Drug: Prevacid

INTERVENTIONS:
Drug: Prevacid — 30mg of Lansoprazole twice daily (or placebo)for eight weeks.

SUMMARY:
The purpose of this study is to determine whether treatment with twice-daily Lansoprazole 30mg (Prevacid 30mg) and behavioral modifications for reflux is superior to treatment with behavioral modifications for reflux alone in the treatment of laryngopharyngeal reflux (LPR).

DETAILED DESCRIPTION:
Laryngopharyngeal reflux (LPR) is a disorder caused by acid-induced damage to the larynx and pharynx (voice box and throat). The standard care for persons with this disorder is treatment with highly potent anti-acid medications (proton pump inhibitors - Prevacid is one of these. NExium, Aciphex and Prilosec are others). These medications are currently approved by the FDA for the treatment of gastroesophageal reflux disease (GERD). Although the use of these medications in persons with LPR is widely accepted and sanctioned, this research is being done because these medications are not currently approved by the FDA for this use. The purpose of this study is to determine whether treatment with twice-daily Lansoprazole 30mg (Prevacid 30mg) and behavioral modifications for reflux is superior to treatment with behavioral modifications for reflux alone in the treatment of laryngopharyngeal reflux (LPR).

ELIGIBILITY:
Inclusion Criteria:

* patients with a clinical diagnosis of laryngopharyngeal reflux diagnosed by any combination of patient symptoms, physical/endoscopic findings, and 24 hr dual-probe ambulatory pH-testing.
* 18 years of age or older

Exclusion Criteria:

* patients with life-threatening complications of laryngeal, pharyngeal or esophageal cancer, subglottic or tracheal stenosis, laryngeal papilloma, airway compromise
* elite vocal performs with LPR-related dysphonia
* under 18 years of age
* pregnant and/or lactating women
* persons with known hypersensitivity to any component of the formulation
* patients taking theophylline, ketoconazole, ampicillin or digoxin
* persons with hepatic and renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2005-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of twice daily Lansoprazole 30mg to placebo in the treatment of laryngopharyngeal reflux symptoms and findings. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Belafsky, MD, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States